CLINICAL TRIAL: NCT01676792
Title: A Pilot Study to Assess the Efficacy & Safety of Topical SR-T100 Gel in the Treatment of Human Vulva Pre-cancerous Lesions (Vulvar Intraepithelial Neoplasia; VIN) & Cutaneous Condyloma(External Genital Warts; EGWs)
Brief Title: SR-T100 Gel Efficacy & Safety Study for Vulva Pre-cancerous Lesions & Cutaneous Condyloma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100CT221; 100CT221 (Other: National Research Program for Biopharmaceuticals, NRPB)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Vulvar Intraepithelial Neoplasia; Genital Warts
Keywords: condyloma acuminate; ano-genital warts; genital warts; cutaneous condyloma; Vulva pre-cancerous lesions; Vulvar Intraepitheral Neoplasia; VIN; EGW
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lesion reduction (Experimental)
  Interventions: Drug: SR-T100 gel with 2.3% of SM in Solanum undatum plant extract

INTERVENTIONS:
Drug: SR-T100 gel with 2.3% of SM in Solanum undatum plant extract — Self administered topical SR-T100 gel on lesion(s) including its peripheral normal skin approximately 1cm around the lesion with the amount of 0.02 g/cm squared with occlusive dressing once daily. Patients who is unable to tolerate with occlusive dressing is instructed 3 times daily in the morning, afternoon & before bed time. Medication should be reapply after bathing or cleaning.
  Other Names: SR-T100 gel

SUMMARY:
This pilot clinical study is to evaluate the efficacy & safety of SR-T100 gel (2.3% of SM in Solanum undatum plant extract) in patients with VIN(s) or EGW(s).

DETAILED DESCRIPTION:
An open-label, pilot study to evaluate the efficacy & safety profiles of SR-T100 gel in treating patients with VINs or EGWs. Male & female older than 20 years old have at least one VIN or EGW with lesion size greater than 5 mm in diameter are candidates for this study. The primary endpoint is evaluated based on patients who has received 16-week treatment and presents evaluable measurement datas by the end of 20th week. The secondary endpoints will be evaluated based on all patients with measurable values for VINs or EGWs, recruited patients in this study has never had experiencs associated with prior SR-T100 treatment of any sorts during their life time before becoming a participant in this study. The study plans to recruit 20 patients with VINs or EGWs, the enrollment duration will last two years with total of 40 patients involved.

ELIGIBILITY:
(EGW group)Inclusion Criteria:

* Male & female patients older than 20 years old presents at least one pathologically confirmed with histopathology EGW with lesion size greater than 5mm in diameter.

(EGW group)Exclusion Criteria:

* Patients with invasive neoplasia, enlarged lymph nodes invasive squamous cell carcinoma, having treated with other investigational drugs within 30 days, pregnancy & lactating females, female with pregnancy potential without using effective boundary barrier or patients with immune-deficience.

(VIN group)Inclusion Criteria:

* Female patients older than 20 years old presents at least one histopathologically confirmed VIN with lesion size greater than 5mm in diameter.

(VIN group)Exclusion Criteria:

* Patients with invasive neoplasia, enlarged lymph nodes invasive squamous cell carcinoma, having treated with other investigational drugs within 30 days, pregnancy & lactating females, female with pregnancy potential without using effective boundary barrier or patients with immune-deficience.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Patients achieve greater than or equal to 75% lesion size reduction | 20 weeks (16 weeks treatment period + 4 weeks follow-up period)
  Proportion of patients achieving greater than or equivalent to 75% lesion size reduction from baseline on the 20th week after 16 weeks of SR-T100 gel treatment

SECONDARY OUTCOMES:
Total clearance rate | 20 weeks (16 weeks treatment period + 4 weeks follow-up period)
  Proportions of patient with treated VIN(s) or EGW(s) completely eradicate.
Partial clearance rate | 20 weeks (16weeks treatment period + 4 weeks follow-up period
  Proportions of patient with treated VIN(s) or EGW(s) size reduction is greater than 75% in volume from baseline.

OTHER OUTCOMES:
Safety | 16 weeks
  To evaluate safety profile of SR-T100 gel by adverse events, serious adverse events, PEs, vital signs & laboratory data changes.

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Fu Hsu, MD, PhD., Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan